CLINICAL TRIAL: NCT03091738
Title: Ramelteon for Treatment of Insomnia in Cirrhosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM13968; 5R01DK087913 (NIH)
Record Dates: First submitted 2017-03-16; First posted 2017-03-27 (Actual); Results first posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Cirrhosis
Keywords: sleep
MeSH Terms: conditions — Fibrosis | interventions — ramelteon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ramelteon Pill (Experimental): Patients given ramelteon and re-evaluated after 15 days of therapy
  Interventions: Drug: Ramelteon Pill

INTERVENTIONS:
Drug: Ramelteon Pill — Patients with compensated cirrhosis and insomnia will be provided ramelteon
  Other Names: Ramelteon

SUMMARY:
To study the effect of ramelteon, a melatonin receptor agonist, on sleep quality, duration and cognitive function in cirrhotics with insomnia.

Patients with cirrhosis have difficulties with their sleep quality, which adversely affects their health-related quality of life. It is assumed the sleep disturbances are related to hepatic encephalopathy (HE) in these patients. However, several recent reports have indicated that this is not a perfect concordance and that cognition is not related to sleep disturbance. The mechanism for this change is not clear, although there is evidence of melatonin-delayed phase in these patients as well as difficulties with the excretion pattern of cortisol. Ghrelin is an orexigenic hormone produced by the stomach which stimulates the appetite and also has a profound effect on sleep. Our group has demonstrated a substantial alteration in ghrelin secretion in cirrhosis that correlates with poor slow-wave sleep. In healthy individuals, ghrelin injection encourages slow-wave sleep while sleep deprivation increases ghrelin levels. The role of ghrelin in the sleep disturbances of cirrhosis has not been determined. Prior studies have also lacked the use of overnight polysomnography as a tool and have relied on either actigraphy or questionnaires. There is a need for detailed mechanistic and therapeutic approaches to analyzing sleep disturbances in cirrhosis.

Also the therapy of sleep disturbance in cirrhosis is largely empirical. Prior studies have evaluated hydroxyzine which runs the risk of precipitating HE. Ramelteon is a melatonin analog that is FDA-approved for use in insomnia and will potentially be useful to restore the sleep-wake cycle in cirrhosis-associated sleep disturbance.

The investigators aim to study the impact of the FDA-approved ramelteon on the sleep quality (using questionnaires and sleep diaries) on these patients with cirrhosis.

DETAILED DESCRIPTION:
This study will be a prospective study of patients with compensated cirrhosis This study will be divided into screening and post-ramelteon visits.

For this study, subjects with cirrhosis will be recruited from the hepatology clinic.

Screening: All subjects will come for an initial screening visit to the CRSU at which point the following procedures will be performed:

1. Vitals, including BMI
2. Neck circumference
3. Skinfold thickness and waist-hip ratio
4. Beck Depression Inventory (BDI)
5. Sickness impact profile for overall HRQOL

Questionnaires regarding sleep:

1. Berlin questionnaire
2. STOP Bang questionnaire
3. Epworth sleepiness scale (ESS) and
4. Pittsburgh sleep quality index (PQSI)

Cirrhotic patients with either of the criteria below (a) neck circumference >17 inches for men and >16 inches for women (b) Positive Berlin questionnaire will be excluded because these are highly suggestive of sleep disturbances and OSA. The investigators will also exclude patients who have evidence of moderate to severe depression on Beck Depression Inventory (score ≥20) without the suicide question.

All enrolled study participants will perform 5 paper-pencil and two computerized tests of intelligence which will last approximately 35 minutes total.

RAMELTEON THERAPY:

The subjects' study chart, current medications, medical history and pregnancy testing will be assessed by sleep physicians at VCU, who will then decide if this patient would benefit from ramelteon.

The criteria used will be insomnia along with the absence of OSA by the questionnaires. Ramelteon is an FDA-approved selective melatonin receptor 1 and 2 analog indicated for use in insomnia. The dose used will be 8 mg, the lowest possible dose. If the sleep specialists believe that a particular cirrhotic patient is a candidate for this therapy, they will be clinically prescribed ramelteon after a detailed face to face visit explaining the risks and benefits. Ramelteon is not indicated in patients with severe hepatic impairment (defined as Child Class C), therefore, these patients will not be included in this study.

If the patient agrees to take the medicine, it will be dispensed through the investigational pharmacy, where it will be stored for this study. Patients will be asked to complete a medication and sleep diary for the duration of the drug therapy which will be a maximum of 15 days. Within 15 days of drug initiation, the patients will be asked to complete the sleep questionnaires again and cognitive testing similar to that described in visit 1.

ELIGIBILITY:
Inclusion Criteria:

* Child class A cirrhosis proven by biopsy, radiology or endoscopic evidence of varices - Able to give informed consent

Exclusion Criteria:

* Patient unwilling to start therapy
* Allergic reactions to ramelteon in the past
* Obstructive sleep apnea
* Periodic limb movement disorder
* Moderate to severe depression
* Unable to give informed consent
* Night shift workers
* Inter-continental travel within the last 4 weeks
* Renal insufficiency on dialysis
* Current alcohol or illicit drug use
* Diabetes Mellitus using insulin therapy
* Use of chronic hypnotic medications more than once per week or more than 5-6 times per month

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jasmohan S Bajaj, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ramelteon Pill
Started | 10
Completed | 8
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ramelteon Pill
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Sleep Quality Evaluation
Description: Pittsburgh Sleep Quality Index (PSQI) is a 19 item survey measuring 7 components of sleep. Component scores are summed to yield a global PSQI score. Scores range from 0 to 21 with higher scores indicate worse sleep quality.
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ramelteon Pill
Number analyzed (Participants) | 8
score on a scale
  Baseline | 4.63 (2.97)
  Day 14 | 11.75 (4.68)

2. Secondary Outcome: Daytime Sleepiness Evaluation
Description: Epworth Sleepiness Scale asks participants to rate (on a scale of 0 to 3) their likelihood of falling asleep during 8 daily activities. Scores range from 0 to 24 with lower scores indicating less sleepiness.
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ramelteon Pill
Number analyzed (Participants) | 8
score on a scale
  Baseline | 4.68 (2.63)
  Day 14 | 5.8 (3.39)

3. Secondary Outcome: Sickness Impact Profile
Description: Sickness Impact Profile is a 68 question assessment. Items are scored 0 (no) or 1 (yes). Scores range from 0 to 68 with higher numbers indicating worse quality of life.
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ramelteon Pill
Number analyzed (Participants) | 8
score on a scale
  Baseline | 4.9 (6.85)
  Day 14 | 3.96 (7.03)

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Ramelteon Pill
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramelteon Pill (N=10)
Paradoxical reaction (Product Issues) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-09-04): https://cdn.clinicaltrials.gov/large-docs/38/NCT03091738/Prot_SAP_001.pdf